CLINICAL TRIAL: NCT03276884
Title: Growth and Tolerance of Young Infants Fed Amino Acid-Based Formulas
Brief Title: Growth and Tolerance of Young Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AL23
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Growth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Infant Formula (Experimental): Infant formula powder to be fed ad libitum
  Interventions: Other: Experimental Infant Formula
- Control Infant Formula (Active Comparator): Infant formula powder to be fed ad libitum
  Interventions: Other: Control Infant Formula

INTERVENTIONS:
Other: Experimental Infant Formula — amino acid-based infant formula powder
  Arms: Experimental Infant Formula
Other: Control Infant Formula — amino acid-based infant formula powder
  Arms: Control Infant Formula

SUMMARY:
To compare growth and tolerance of healthy term infants fed two amino acid-based infant formulas.

ELIGIBILITY:
Inclusion Criteria:

* Subject is judged to be in good health.
* Singleton from a full-term birth with a gestational age of 37 - 42 weeks.
* Birth weight was ≥ 2490 g (~5 lbs. 8 oz.).
* Subject is between 0 and 8 days of age at enrollment.
* Parent(s) confirm their intention to feed their infant the study product as the sole source of nutrition for the duration of the study.
* Parent(s) confirm their intention not to administer vitamin or mineral supplements (with the exception of Vitamin D-containing supplements), solid foods or juices to their infant from enrollment through the duration of the study.
* Subject's parent(s) has voluntarily signed and dated an ICF prior to any participation in the study.

Exclusion Criteria:

* An adverse maternal, fetal or subject medical history that is thought by the investigator to have potential for effects on tolerance, growth, and/or development.
* Subject is taking and plans to continue medications, home remedies, herbal preparations, prebiotics, probiotics or rehydration fluids that might affect gastrointestinal (GI) tolerance.
* Subject participates in another study that has not been approved as a concomitant study.

Max Age: 8 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 267 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Weight Gain | Study Day 14 to Study Day 119
  Infant scale

SECONDARY OUTCOMES:
GI tolerance | Study Day 1 to Study Day 119
  Parent completed questionnaires
Length | Study Day 1 to Study Day 119
  Length board
Head Circumference | Study Day 1 to Study Day 119
  Measure tape
Weight | Study Day 1 to Study Day 119
  Infant scale

CONTACTS AND LOCATIONS:
Overall Officials: Jan Kajzer, MS, RD, LD, Study Chair — Abbott Nutrition
Locations (22):
- United States (22):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Southeastern Pediatric Associates, Dothan, Alabama
  - Watching Over Mothers and Babies, Tucson, Arizona
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - Norwich Pediatric Group, PC, Norwich, Connecticut
  - Children's Research, LLC, Lake Mary, Florida
  - Score Physician Alliance, LLC, St. Petersburg, Florida
  - Saltzer Medical Group, Nampa, Idaho
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Springs Medical Research, Owensboro, Kentucky
  - Women's Clinic of Lincoln, PC, Lincoln, Nebraska
  - Pediatric Associates of Fairfield, Inc., Fairfield, Ohio
  - Institute of Clinical Research, LLC, Mentor, Ohio
  - The Cleveland Pediatric Research Center, LLC, Middleburg Heights, Ohio
  - Medical Research South, Charleston, South Carolina
  - Coastal Pediatric Research 3002, Charleston, South Carolina
  - Coastal Pediatric Associates 3004, Mt. Pleasant, South Carolina
  - Coastal Pediatric Research 3003, North Charleston, South Carolina
  - Memphis & Shelby County Pediatric Group, Memphis, Tennessee
  - Vilo Research Group Inc, Houston, Texas
  - Southwest Children's Research Associates, PA, San Antonio, Texas
  - Tanner Clinic, Layton, Utah

IPD SHARING:
Plan to Share IPD: Undecided